CLINICAL TRIAL: NCT06901128
Title: The Covideo Study - a Randomized Controlled Trial of Cognitive Therapy for Social Anxiety Disorder in Youth, Comparing Screen to Office Delivery
Brief Title: The Covideo Study - a Trial of Cognitive Therapy for Social Anxiety Disorder in Youth, Comparing Screen to Office Delivery
Acronym: Covideo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Helse Vest (Other); University of Oslo (Other); St. Olavs Hospital (Other); University of Oxford (Other); University of Bergen (Other); Norwegian University of Science and Technology (Other); University of Tromso (Other); Yale University (Other); Linkoeping University (Other Government); University of Aarhus (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18736585; 2022209 (Other Grant/Funding Number: Nasjonalt program for klinisk behandlingsforskning i spesialisthelsetjenesten KLINBEFORSK. Grant Number 2022209.)
Record Dates: First submitted 2025-02-28; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: RCT video screen delivery cognitive therapy youth
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screen delivery (Experimental): CT by video/screen
  Interventions: Behavioral: cognitive therapy
- Office delivery (Active Comparator)
  Interventions: Behavioral: cognitive therapy

INTERVENTIONS:
Behavioral: cognitive therapy — The CT-SAD-A manual developed by Clark and Leigh

SUMMARY:
The main goal of this clinical trial is to examine screen delivery as an alternative for offering cognitive therapy to youth with social anxiety. It will examine its effectiveness compared to office delivery, but also its acceptability and sustainability, and identify factors important for the outcome of this approach.

The main questions it aims to answer are:

Does screen delivery show comparable effectiveness to office delivery? Is screen delivery well accepted by youth and therapists? Does screen delivery show economic and climate sustainability? Do credibility and therapeutic alliance predict therapy outcome?

In the study researchers will compare screen delivery to office delivery of cognitive therapy for social anxiety disorders in 200 youth aged 14-18 years.

After an initial screening in schools, eligible youth are assessed with a diagnostic interview. Those meeting inclusion criteria will be offered either screen or office therapy. This is decided by random selection (a draw).

Participants will:

Complete an initial short screening questionnaire. Respond to a diagnostic interview online. Meet their therapist first time in person. Attend 14 weekly 90-minutes therapy session. Complete weekly questionnaires during the therapy. Answer interview and questionnaires after the therapy, and also 6 months, 2 years and 4 years later. Parents are also interviewed and informed of the study.

DETAILED DESCRIPTION:
Study aim The main aim of the study is to evaluate screen delivery (SD) as an alternative approach to traditional office delivery (OD) for reaching young people with cognitive therapy (CT) for Social Anxiety Disorder (SAD). In this multi-centre randomized controlled trial (RCT) includes three work packages (WPs), focusing on effectiveness (WP1), acceptability (WP2), health economy and sustainability (WP3), and predictors for outcome (WP4). We aim to show that effectiveness of CT for SD is not inferior compared to OD, that CD is well accepted by youths and therapists, that CD has economic and climate benefits over OD, and we will identify predictors for therapy outcome. SD may represent a novel way of increasing access to effective therapy for young people, leading to improved health and success in education, employment and social life.

Screen delivery (SD) The study originates from the Child and Adolescent Mental Health Services (CAMHS) department at Innlandet Hospital, Norway. Innlandet CAMHS covers a large and mainly rural area, with some clients having long travel distances, and with very limited public transportation. Video communication with patients and families has therefore been of interest to our department over the last decade.

Early into the Covid-19 pandemic, a survey among clinicians in our department found high satisfaction with consultations on screen, especially among younger clinicians (below 40 years of age), and in the treatment of anxiety disorders (after an initial office consultation). A subsequent paper confirmed and extended our findings, noting several potential advantages for SD over OD, including time and cost for travel, logistics, inclusion of "hard to reach" family members, and the possibility to observe clients in their natural setting. This inspired the present study where we examine SD for anxiety in youth.

Public demand and state of the art In 2001 the Norwegian government set a target for at least 15% virtual consultations within the specialist health service. The following year, our four regional health authorities launched a plan for 40% reduction in CO2e-emission by 2030, stating that 20% of consultations should be by screen or telephone. Being the closest analogue to OD, SD may have the potential to reach out to people with effective, acceptable and sustainable mental health interventions. Following more than three decades of research, several online therapy manuals have acquired a solid evidence base. Contrasting this, surprisingly little has been published on SD, especially in light of the surge in its use after the pandemic. Two recent reviews of SD of mental health interventions identified only a single pilot study with adolescents. A review of SD in cognitive behavior therapy (CBT) needed to exclude youth due to lack of studies, urging future original studies to include this age group.

Social Anxiety Disorder SAD is prevalent, with a life-time prevalence around 13%, and a median age of onset of 13 years. Untreated, it follows a chronic course throughout the lifespan, with adverse effects on mental health, education, employment, social life and family life. Treatment is often delayed for years or decades, until those affected develop comorbid depression or substance abuse, and/or drop out of education or work. Social isolation and unstable family life are frequent consequences. Early and easy access to effective treatment is therefore important to prevent such negative impact on mental health and development, and also to reduce school absenteeism in youth which has risen sharply after the pandemic.

CT for SAD Members of our consortium have been involved anxiety treatment studies for decades. In Norway, generic CBT programs for common child anxiety disorders (SAD, separation anxiety disorder and generalized anxiety disorder), are usually offered at CAMHS. However, our studies documented lower recovery for SAD compared to the other two common anxiety disorders, a finding since confirmed in a recent review and meta-analysis by other members of our consortium. Already three decades ago, a CT manual, specifically for adults with SAD, was developed by a member of our consortium. It has subsequently shown excellent effect in a long range of studies. Another of our members also found this manual effective in youth, when delivered individually at the office in CAMHS. Recently, an official adaptation of the manual was developed for adolescents (named CT-SAD-A). Initial studies of office and online delivery of the manual showed promising results, and was therefore selected as the intervention for this study where we aim to compare SD to OD in the treatment of SAD in youth.

Study design The study is an RCT with two-arms and a non-inferiority design. Youth are randomized 1:1 to the two delivery modes, stratified by therapist. Planned inclusion period is 3 years.

Recruitment and screening We will recruit youth referred to Child and Adolescent Mental Health Services (CAMHS) and youth seeking municipal services, as well as youth identified by screening at high-schools with an established three-item SAD symptom questionnaire, the Mini-SPIN. Local coordinators will oversee screening and recruitment at the study sites.

Intervention Therapy sessions with the CT-SAD-A will be delivered weekly for 14 weeks, each with a 90-minutes duration. A booster session is offered 6-months post treatment.

Feasibility A feasibility study, involving focus group interviews and questionnaires with completed by 15-20 therapists, and questionnaires completed by a similar number of youth and parents, will be conducted at the start of the study.

Therapists and clinics Therapists are recruited both from CAMHS and municipal health services at four regional sites: Helse SørØst, else Vest, Helse Midt and Helse Nord.

Members of our consortium who developed the CT-SAD-A manual will provide therapist training. In the pilot stage therapists are required to treat one youth with SAD by SD and one by OD, while attending weekly group supervision. Study sites are established in all four Norwegian health regions.

Data storage and handling The Microsoft video system Teams is used for recording and storage from all therapy sessions, as well as interview data. Questionnaire data collected online is stored by use of CheckWare; a system approved in all health regions. Therapists are automatically informed when questionnaires have been completed, and if responses indicate any serious concern, having immediate access to all responses.

Data quality A random 15% of therapy sessions (n=420) will be extracted and examined for adherence to the therapy manual and therapeutic competence, using a purpose-made standardized measure.

Statistical analyses The primary population will be the per-protocol population, with additional sensitivity analyses on the intention-to-treat population. The primary outcome will be analyzed in a mixed model framework, accounting for stratification factors and confounders. Power was calculated for the primary outcome measure, the Liebowitz Social Anxiety Scale Children/Adolescents self-report version (LSAS-CA), with noninferiority design, and 1:1 patient allocation. Non-inferiority margin was set at 10, with a standard deviation of 18. With these assumptions, and a confidence level of 95%, a sample of 144 subjects will result in 95% power. Inclusion of 200 youth allows for an estimated 20% pre to post attrition and 10% post to booster attrition.

Therapist number With 20 therapists treating two patients per semester in year one, and three patients per semester in year two, 200 patients will receive treatment within the planned inclusion period. Inclusion of therapists and patients will go on until inclusion is complete. Training seminars for new therapists on the manual and technical procedures will be conducted regularly.

Risk management Risk to participants is considered minimal. Significant distress during treatment has not occurred in previous case series, or in the pilot stage. Close collaboration with parents is maintained throughout the study. Weekly reports on anxiety and depression are collected, and signs of deterioration noticed by therapists. An item for suicidality is added to the Short Mood and Feelings Questionnaire (SMFQ), item 19 from its long version. Any report of this is or any other sign of deterioration or elevated risk will promptly be acted upon with appropriate procedures and additional or alternative treatment offered when appropriate.

Necessary equipment Youth will use their own smartphones, tablets or personal computers, both for SD sessions and for completion of questionnaires. Clinicians are provided with laptops and web-cameras.

Budget and funding Total cost incl. self-financing was estimated at NOK 39,884 million for the duration of the study, but training of therapists and therapy delivery also in the municipalities will involve additional study costs. The main funding of NOK 18,379 million comes from a National program for clinical treatment research (Klinbeforsk), organized by the regional health authorities of Norway. Running costs for the study, as well as funding for one PhD student, and a PostDoc position, and research assistants, is covered by this grant. One PhD and running costs for the pilot stage is funded by Innlandet Hospital Trust (the sponsor), while the one PhD is co-funded by Innlandet Hospital and the Regional Health Authority for South/Eastern Norway.

Plan for activities, visibility, and dissemination During the pilot stage that started in February 2022, training seminars with therapists have been conducted, and weekly group therapy supervision has been provided. The first training seminars was recorded for use with new therapists coming into the study later. A 3 year inclusion period is planned from February 2025, with 2- and 4-year post-treatment follow-ups. We expect four PhDs and the PostDoc to produce at least 15-20 original papers from the study, which we aim to publish in high-ranking international peer-reviewed open-access journals. Findings will also be presented at conferences, to patients, the health service, and authorities.

Plan for implementation Implementation of SD as a delivery mode in CAMHS and municipalities is ongoing. Data on effectiveness, acceptability, and sustainability will speed up this process. Clinicians from the study will contribute to local implementation, and SD training throughout Norway will be arranged when the study has provided positive results. The CT-SAD-A manual will also be made available to services in all four health regions. Presentations at national and international conferences, meetings and seminars, as well as dissemination through user organizations, will also be important for implementation.

User involvement A user representative from the Youth Council at Innlandet Hospital has been recruited, taking part in planning and development of information and consent letters, interview guides and questionnaires, and will contribute in dissemination to youth, the public and government.

Ethical considerations The study is approved by the Regional Committee for Medical and Health Research Ethics, and by the Data Protection Officer at Innlandet Hospital Trust. The study involves children, and informed assent (below 16 years) or consent from youth and parents is required. Participants may withdraw at any time without negative consequences. Additional or alternative therapy will be offered in case of deterioration or insufficient effect.

ELIGIBILITY:
Inclusion Criteria:

* Social anxiety disorder primary
* Age 14 to 18 years.
* Norwegian fluency

Exclusion Criteria:

* Severe Depression
* Acute suicidality
* Substance abuse
* Psychosis
* Intellectual Disability
* More than 20% absence from school in previous three months

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Liebowitz social anxiety scale for children and adolescents (LSAS-CA) | From start of treatment until end of 14 weekly treatment sessions.
  24 item scale rated in four response categories
Anxiety and Related Disorders Interview Schedule for DSM-5 Chid and parent Version | From start of treatment until end of 14 weekly treatment sessions.
  Short name ADIS-5 C/P.

SECONDARY OUTCOMES:
Revised Children´s Anxiety and Depression Scale RCADS | From start of treatment until end of 14 weekly treatment sessions.
  Symptom measure for anxiety and depression in children
Short Mood and Feelings Questionnaire SMFQ | From start of treatment until end of 14 weekly treatment sessions.
  Symptom measure for anxiety and depression for youth
Strengths and Difficulties Questionnaire SDQ | From start of treatment until end of 14 weekly treatment sessions.
  Screening measure for mental disorders in youth

CONTACTS AND LOCATIONS:
Overall Officials: Einar R Heiervang, MD PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (5):
- Norway (5):
  - Sykehuset Innlandet, Forskningsavdelingen, Sanderud Sykehus, Ottestad, Innlandet
  - Helse Vest, Førde
  - Helse SørØst, Hamar
  - Helse Nord, Tromsø
  - Helse Midt, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
IPD for all participants will be shared anonymously with other researchers following reasonable requests.
Supporting Information: Study Protocol, ICF
Time Frame: February 10, 2025 - December 31, 2035
Access Criteria: Access to the above provided following information for use provided to the PI.

REFERENCES:
- [Background] Leigh E, Clark DM. Understanding Social Anxiety Disorder in Adolescents and Improving Treatment Outcomes: Applying the Cognitive Model of Clark and Wells (1995). Clin Child Fam Psychol Rev. 2018 Sep;21(3):388-414. doi: 10.1007/s10567-018-0258-5. PMID 29654442